CLINICAL TRIAL: NCT00700908
Title: The Impact of an Automated Telephone Intervention on HbA1c in Type 2 Diabetes: A Randomized Controlled Trial
Brief Title: Impact of an Automated Telephone Intervention on Glycosylated Hemoglobin (HbA1c) in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0701M99406
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; telephone intervention; automated
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Automated telephone intervention
  Interventions: Behavioral: automated telephone intervention vs. usual care
- 2 (Active Comparator): Usual care
  Interventions: Behavioral: automated telephone intervention vs. usual care

INTERVENTIONS:
Behavioral: automated telephone intervention vs. usual care

SUMMARY:
Aim 1. Determine the impact of a daily, automated telephone intervention on HbA1c levels compared to standard care in older patients with type 2 diabetes.

Aim 2. Determine the impact of the automated telephone intervention compared to standard care on adherence to prescribed SMBG frequency in older patients with type 2 diabetes.

Aim 3. Determine the impact of the automated telephone intervention compared to standard care on self-reported diabetic control problems in older patients with type 2 diabetes.

Aim 4. Determine the impact of the automated telephone intervention compared to standard care on self-reported attitudes and health beliefs concerning diabetes in older patients with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* Age greater or equal to 55
* Type 2 diabetes
* English speaking
* Ability to use glucose meter

Exclusion Criteria:

* Unable to give informed consent
* Unwilling to allow SMBG levels to be shard with primary care physician

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | three months

SECONDARY OUTCOMES:
Change in adherence to SMBG frequency | three months

CONTACTS AND LOCATIONS:
Overall Officials: Judith Graziano, PhD, RN, Principal Investigator — University of Minnesota
Locations (1):
- Primary Care Center University of Minnesota, Minneapolis, Minnesota, United States